CLINICAL TRIAL: NCT05881746
Title: Anatomical Resection Versus Nonanatomical Resection for Colorectal Liver Metastases Patients With Gene Mutation or Right-sidedness: The ARCLAMP Randomized Controlled Trial
Brief Title: Anatomical Resection VS. Nonanatomical Resection for Colorectal Liver Metastases With Gene Mutation or Right-sidedness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Director of the Department of Colorectal Surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARCLAMP
Record Dates: First submitted 2023-05-15; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Carcinoma; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anatomical resection group (Experimental): Based upon the segmental anatomy of the liver according to Couinaud system, anatomical resection (AR) is defined as the resection of one or more complete hepatic segments in our study, including bisegmentectomy, right hemihepatectomy, left hemihepatectomy, extended right hemihepatectomy, extended left hemihepatectomy, single segmentectomy, caudate lobectomy, or a combination thereof.
  Interventions: Procedure: anatomical liver resection
- nonanatomical resection group (Active Comparator): nonanatomical resection (NAR), also called as wedge resection, is defined as the resection of the tumor with a margin of normal parenchyma regardless of the hepatic anatomy.
  Interventions: Procedure: nonanatomical liver resection

INTERVENTIONS:
Procedure: anatomical liver resection — Based upon the segmental anatomy of the liver according to Couinaud system, anatomical resection (AR) was defined as resection of 1 or more complete hepatic segments in our study, including bisegmentectomy, right hemihepatectomy, left hemihepatectomy, extended right hemihepatectomy, extended left hemihepatectomy, single segmentectomy, caudate lobectomy, or a combination of these.
  Arms: anatomical resection group
Procedure: nonanatomical liver resection — Nonanatomical resection(NAR), known as wedge resection, was defined as resection of the tumor with a margin of normal parenchyma without regard to hepatic anatomy.
  Arms: nonanatomical resection group

SUMMARY:
In this study, colorectal cancer patients with initially resectable liver-only metastases, as prospectively confirmed by a local multidisciplinary team (MDT) according to predefined criteria, will be tested for RAS and BRAF tumor mutation status. Patients with gene mutant or right-sidedness will be randomised between anatomical resection (AR) or nonanatomical resection (NAR). The primary end-point is the relapse-free survival.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized control trial. The major including criteria are (1) Histologically confirmed colorectal cancer initially resectable liver-only metastases ; (2) patient has the opportunity to perform either anatomical resection (AR) or nonanatomical resection (NAR) surgery; (3) the number of metastasis is 1-3; (4) KRAS/NRAS/BRAF mutation or right-sidedness. Patients will be randomised between AR or NAR. Patients will be stratified for gene mutation and right-sidedness.

Based upon the segmental anatomy of the liver according to Couinaud system, AR is defined as the resection of one or more complete hepatic segments in our study, including bisegmentectomy, right hemihepatectomy, left hemihepatectomy, extended right hemihepatectomy, extended left hemihepatectomy, single segmentectomy, caudate lobectomy, or a combination thereof. NAR, also called as wedge resection, is defined as the resection of the tumor with a margin of normal parenchyma regardless of the hepatic anatomy.

The primary end-point is the relapse-free survival. The secondary end-points are postoperative complication, postoperative mortality, hospital length of stay, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years;
2. Histological proof of colorectal adenocarcinoma;
3. Resectable colorectal liver metastasis without detectable extrahepatic distant metastatic disease (determined by a local MDT);
4. Suitable for anatomical or nonanatomical liver resection (determined by a local MDT);
5. Number of metastasis is 1 to 3;
6. KRAS/NRAS/BRAF mutation or right-sidedness;
7. Performance Status (ECOG) 0~1;
8. Adequate hematological function: Neutrophils≥1.5 x109/l and platelet count≥100 x109/l; Hb ≥9g/dl (within 1 week prior to randomization);
9. Adequate liver and renal function: total bilirubin ≤2.0 mg/dl, serum transaminases ≤ 5x upper limit of normal(ULN), and serum creatinine ≤ 1.5x ULN and creatinine clearance ≥ 30 ml/min;
10. Written informed consent.

Exclusion Criteria:

1. Previous systemic treatment for metastatic disease;
2. Previous surgery for metastatic disease;
3. Extrahepatic metastases;
4. Unresectable primary tumor;
5. Major cardiovascular events (myocardial infarction, severe/unstable angina, congestive heart failure, CVA) within 12 months before randomisation;
6. Second primary malignancy within the past 5 years;
7. Acute or subacute intestinal obstruction;
8. Drug or alcohol abuse;
9. No legal capacity or limited legal capacity;
10. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
relapse-free survival | 3 years
  The relapse-free survival (PFS) was defined as the period from the start of initial liver resection to the date of tumor relapse or death

SECONDARY OUTCOMES:
overall survival | 5 years
  The overall survival (OS) was defined as the period from the start of initial liver resection until death from any cause, at which point the data was censored.
postoperative hospital stay | 30 days post operatively
  The postoperative hospital stay is defined as the number of date from the first day after operation to discharge.
postoperative complication | After surgery during one month
  Patients will be evaluated for surgical morbidity during 1 month. Postoperative morbidity will be scored according 'Clavien-Dindo Grade'.
postoperative mortality | After surgery during 90 days
  any death occured within 90 days after the last resection of primary and metastatic lesions

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No